CLINICAL TRIAL: NCT02116426
Title: The Role of Copeptin Testing During Pre-hospital Care in the Treatment of Chest Pain Suggestive of Acute Coronary Syndrome
Brief Title: Copeptin Testing During Pre-hospital Care in the Treatment of Chest Pain Suggestive of Acute Coronary Syndrome
Acronym: SCA COP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2013/PGC-01; 2013-A01201-44 (Other: RCB number:)
Record Dates: First submitted 2014-04-15; First posted 2014-04-16 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Chest Pain
Keywords: copeptin; troponin HS
MeSH Terms: conditions — Chest Pain; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- The study population: The study population includes all adult patients taken in charge by the emergency ambulance services of the participating centers for non-traumatic chest pain for suspected Acute Coronary Syndrome (ACS) without ST segment elevation.
  Intervention: Blood work in the ambulance Intervention: Blood work upon arrival in the emergency room Intervention: Blood work at 3 hours post-arrival in the emergency room
  Interventions: Biological: Blood work in the ambulance; Biological: Blood work upon arrival in the emergency room; Biological: Blood work at 3 hours post-arrival in the emergency room

INTERVENTIONS:
Biological: Blood work in the ambulance — Blood sample for copeptin and troponin HS testing is taken during ambulance care.
Biological: Blood work upon arrival in the emergency room — Blood in drawn for copeptin and troponin HS testing upon arrival in the emergency room.
Biological: Blood work at 3 hours post-arrival in the emergency room — Blood is drawn for troponin HS testing 3 hours after the patient's arrival in the emergency room.

SUMMARY:
The main objective of our study is to evaluate the diagnostic value of copeptin testing in association with troponin HS testing during pre-hospital care (ambulance care) in the treatment of patients whose pattern of use is the occurrence chest pain suggestive of ACS but not ST+.

DETAILED DESCRIPTION:
The secondary objectives of this study are to:

A. Evaluate the diagnostic value of determination of copeptin testing in pre-hospital care in another diagnosis;

B. Assess the prognostic value of copeptin assay on vital prognosis at day 28;

C. Evaluate the kinetics of copeptin and troponin HS between initial ambulance care and arrival at the emergency department;

D. Evaluate the potential impact of copeptin testing on pre-hospital patient care;

E. Assess the economic impact of pre-hospital copeptin testing in terms of hospital stays and optimizing ambulance movements.

ELIGIBILITY:
Inclusion Criteria:

* all major adult patients taken in charge by the emergency ambulance services of the participating centers for non-traumatic chest pain for suspected ACS and an electrocardiogram initially excluding an ST segment elevation

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient (or a legal representative) formalizes his/her opposition for the study
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* The patient has a contraindication for a treatment used in this study
* The patient's initial electrocardiogram indicates an ST segment elevation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes all adult patients taken in charge by the emergency ambulance services of the participating centers for non-traumatic chest pain for suspected Acute Coronary Syndrome (ACS) without ST segment elevation.
Sampling Method: Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2015-07-29 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Blood troponin HS concentration (µg/L) | Day 0, in the ambulance
Blood copeptin concentration (pmol/l) | Day 0, in the ambulance
Final diagnosis of ACS non ST + (yes/no) | Day 28

SECONDARY OUTCOMES:
Blood troponin HS concentration (µg/L) | Day 0, upon arrival in the emergency department
Blood troponin HS concentration (µg/L) | Day 0, 3 hours after arrival in the emergency department
Mortality | Day 28
Would you leave the patient at home if both copeptin and troponin tests were negative? | Day O (in the ambulance)
  Yes/no question asked of ambulance doctors.
Hospital costs (€) associated with avoidable services | Day 28
Distance (km) between the hospital and the patient's place of residence | Day 28
Time spent by ambulance staff at the patient's place of residence | Day 0
Presence/absence of another diagnosis | Day 28
Number of patients taken in charge that day by ambulance staff. | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Géraud Claret, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CHRU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes